CLINICAL TRIAL: NCT02396953
Title: Phase IIa, Open Label, Dose Ascending Study to Determine the Maximum Tolerated Dose, Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of Lanreotide PRF in Subjects With Acromegaly Previously Treated and Controlled With Either Octreotide LAR or Lanreotide Autogel
Brief Title: Study to Determine the Maximum Tolerated Dose, Safety and Tolerability of a Single Dose of Lanreotide Prolonged Release Formulation (PRF) in Subjects With Acromegaly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-55-52030-309; 2014-002389-62 (EudraCT Number)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lanreotide PRF (Experimental): One single dose of lanreotide PRF (via subcutaneous injection) either 180mg or 270mg or 360mg.
  Interventions: Drug: Lanreotide PRF

INTERVENTIONS:
Drug: Lanreotide PRF
  Other Names: Lanreotide acetate

SUMMARY:
The objectives of the protocol is to determine the maximum tolerated dose and to investigate the pharmacokinetics of a single dose of lanreotide PRF in subjects with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of acromegaly.
* Provided written informed consent prior to any study related procedures.
* Between 18 and 75 years of age inclusive.
* Female of non-childbearing potential or male. Non-childbearing potential is defined as being postmenopausal for at least 1 year, or women with documented infertility (natural or acquired).
* Male subjects must agree that, if their partner is at risk of becoming pregnant, they will use a medically accepted, effective method of contraception (i.e. condom) for the duration of the study (maximum of 7.5 months).
* Treatment with a stable dose of either octreotide LAR or lanreotide Autogel for at least 3 months immediately prior to study entry, with confirmation of disease control during this treatment period (documentation of age adjusted IGF 1 <1.3 x upper limit of normal (ULN), based on local laboratory results, during screening period).
* If the subject is receiving treatment for hypertension, the dose has been stable for at least 1 month prior to study entry.
* Subjects must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow up evaluation as specified in the protocol.

Exclusion Criteria:

* Has undergone radiotherapy within 2 years prior to study entry.
* Has been treated with a dopamine agonist and/or GH receptor antagonist or has undergone pituitary surgery within 3 months prior to study entry.
* Is anticipated to require pituitary surgery or radiotherapy during the study.
* Has clinically significant hepatic abnormalities and/or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥3 x ULN and/or alkaline phosphatase (AP) ≥2.5 x ULN and/or total bilirubin ≥1.5 x ULN and/or gamma-glutamyl transpeptidase (GGT) ≥2.5 x ULN during the Screening period (central laboratory results) or a history of these findings when on somatostatin analogue (SSTa) treatment.
* Has clinically significant pancreatic abnormalities and/or amylase and/or lipase ≥1.5 x ULN during the Screening period (central laboratory results).
* Has any significant renal abnormalities and/or creatinine ≥1.5 x ULN during the screening period (central laboratory results).
* Has uncontrolled diabetes (glycosylated haemoglobin (HbA1c) ≥9%, centrally assessed during the Screening period), or has diabetes treated with insulin for less than 6 months prior to study entry.
* Has any known uncontrolled cardiovascular disease or had any of the following within 6 months of Screening: ventricular or atrial dysrhythmia

  ≥grade 2, bradycardia ≥grade 2, electrocardiogram (ECG) QT interval corrected (QTc) prolonged ≥grade 2, myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, hypertension not adequately controlled by current medications.
* Use of any hormone replacement therapy (HRT) with oestrogens.
* Has symptomatic gallstones/ sludge at the Screening Visit echography (local assessment) OR is asymptomatic but has echography showing clear evidence of impending inflammation such as localised mucosal thickening suggesting the subject is at high risk of developing acute disease. Subjects with asymptomatic gallstones/ sludge and otherwise normal echography may be entered at the discretion of the investigator.
* Has abnormal findings during the Screening period, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety.
* Has been treated with any other investigational medicinal product (IMP) prior to the first study visit without undergoing a washout period of seven times the elimination half-life of the investigational compound.
* Has a known hypersensitivity to any of the test materials or related compounds.
* Is likely to require treatment during the study with drugs that are not permitted by the study protocol.
* Has a history of, or known current, problems with alcohol or drug abuse.
* Has any mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (36):
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Domaine Universitaire Sart Tilman, Liège
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultní nemocnice Hradec Králové (University Hospital Hradec), Hradec Králové
- France (4):
  - CHU le BOCAGE, Dijon
  - Hôpital de Bicêtre (AP-HP), Le Kremlin-Bicêtre
  - CHU de la Timone, Marseille
  - Hôpital Haut Lévêque, Pessac
- Germany (2):
  - University Medicine Berlin, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg
- Italy (6):
  - IRCCS AOU San Martino-IST, University of Genova, Genova
  - Azienda Ospedaliera Padova, Padua
  - Policlinico of Palermo, Palermo
  - Ospedale Cisanello, Pisa
  - Azienda Ospedaliera Universitaria Senese, Siena
  - AO Città della Salute e della Scienza di Torino, Torino
- Lithuania (2):
  - Lithuanian University of Health Sciences (LUHS) Kauno klinikos, Kaunas
  - Vilnius University hospital Santariskiu Klinikos, Vilnius
- Erasmus University Medical Centre Rotterdam, Rotterdam, Netherlands
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Szpital Kliniczny im. H. Święcickiego UM w Poznaniu, Poznan
  - Szpital Bielanski im. ks. Jerzego Popieluszki SPZOZ, Warsaw
  - Szpital Kliniczny nr 1, Wroclaw
- National Institute of Endocrinology, Bucharest, Romania
- Russia (6):
  - Kazan state Medical Academy, Kazan'
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Endocrinological Research Center Ministry of Health Russian Federation, Moscow
  - Healthcare Institution, Nizhny Novgorod
  - Federal State Budgetary Military, Saint Petersburg
  - North-Western State Medical University, Saint Petersburg
- Spain (3):
  - Hospital Universitario Vall d' Hebron, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (3):
  - Queen Mary, University of London, London
  - Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Neggers S, Badiu C, Biagetti B, Durand-Gasselin L, Petit A, Petrossians P, Regnault B, Rich D, Shafigullina Z, Shustov S, Vydrych A. Pharmacological and safety profile of a prolonged-release lanreotide formulation in acromegaly. Expert Rev Clin Pharmacol. 2021 Dec;14(12):1551-1560. doi: 10.1080/17512433.2021.1986004. Epub 2021 Nov 8. PMID 34664531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, dose-ascending study to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability of a single dose of lanreotide prolonged release formulation (PRF). 17 centres recruited adult subjects with acromegaly into 3 lanreotide PRF treatment cohorts (180 milligrams [mg], 270 mg and 360 mg).
Pre-assignment Details: Screening of subjects took place 28 to 42 days before administration of study treatment (Day -42 to Day -28). Overall, 60 subjects were screened during this run-in period; 32 of whom were screening failures and 28 subjects were enrolled and treated with lanreotide PRF.
Groups:
- 180 mg Lanreotide PRF: On Day 1, 3 initial subjects in Cohort 1 received 180 mg lanreotide PRF by a single deep subcutaneous injection in the superior, external quadrant of the buttock and a 12-week treatment period then commenced. The dose escalation proceeded with a 3+3+3 scheme. If 0 or 1 out of the 3 dosed subjects had experienced a dose limiting toxicity (DLT), 3 more subjects would have been dosed with the same dose. If more than 3 out of 9 subjects had experienced a DLT, dose escalation would have been stopped and the dose declared the maximum administered dose. If ≤3 DLTs had been observed in the 9 treated subjects and the overall safety was in line with the known lanreotide safety profile, the data review committee (DRC) would have allowed the dose to be escalated to 270 mg (Cohort 2).
  At the end of the treatment period subjects continued to be assessed over a 12-week follow up period until end of study (EOS) at Week 25 or early withdrawal (EW).
- 270 mg Lanreotide PRF: On Day 1, 1 initial subject in Cohort 2 received 270 mg lanreotide PRF by a single deep subcutaneous injection in the superior, external quadrant of the buttock and a 12-week treatment period then commenced. Cohort 2 subjects were treated and reviewed on a 1+2+2+2+2 scheme. If no DLT was experienced, 2 more subjects would have been dosed with the same dose. If more than 3 out of 9 subjects had experienced a DLT, dose escalation would have stopped, and the dose was declared the maximum administered dose. If ≤3 DLTs had been observed in the 9 treated subjects and the overall safety was in line with the known lanreotide safety profile, the DRC would have allowed dose to be escalated to 360 mg (Cohort 3).
  At the end of the treatment period subjects continued to be assessed over a 12-week follow up period until EOS at Week 25 or EW.
- 360 mg Lanreotide PRF: On Day 1, 2 initial subjects in Cohort 3 received 360 mg lanreotide PRF by a single deep subcutaneous injection in the superior, external quadrant of the buttock and a 12-week treatment period then commenced. Cohort 3 subjects were treated and reviewed on a 2+2+2+3 scheme. An additional subject was also dosed in this cohort as it was considered unethical to exclude an eligible subject. If 0 or 1 subject had experienced a DLT, 2 more subjects would have been dosed with the same dose. If more than 3 out of 9 subjects had experienced a DLT, dose escalation would have been stopped and the dose was declared the maximum administered dose.
  At the end of the treatment period subjects continued to be assessed over a 12-week follow up period until EOS at Week 25 or EW.
Period: Overall Study
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Started | 9 | 9 | 10
Completed | 5 | 6 | 7
Not Completed | 4 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Insulin like Growth Factor-1 increased | 3 | 2 | 2
Not completed — Personal Reasons | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 180 mg Lanreotide PRF: On Day 1, 3 initial subjects in Cohort 1 received 180 mg lanreotide PRF by a single deep subcutaneous injection in the superior, external quadrant of the buttock and a 12-week treatment period then commenced. The dose escalation proceeded with a 3+3+3 scheme. If 0 or 1 out of the 3 dosed subjects had experienced a DLT, 3 more subjects would have been dosed with the same dose. If more than 3 out of 9 subjects had experienced a DLT, dose escalation would have stopped, and the dose declared the maximum administered dose. If ≤3 DLTs had been observed in the 9 treated subjects and the overall safety was in line with the known lanreotide safety profile, the DRC would have allowed the dose to be escalated to 270 mg (Cohort 2).
  At the end of the treatment period subjects continued to be assessed over a 12-week follow up period until EOS at Week 25 or EW.
- Total: Total of all reporting groups
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF | Total
Number analyzed (Participants) | 9 | 9 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 7 | 24
  >=65 years | 1 | 0 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (7.2) | 52.1 (8.7) | 56.2 (11.6) | 55.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 15
  Male | 3 | 4 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 9 | 10 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Prior Acromegaly Medication [Count of Participants; unit: Participants]
  Octreotide Long Acting Release (LAR) | 9 | 7 | 7 | 23
  Lanreotide Autogel | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) by Number of Subjects With DLTs.
Description: The MTD was defined based on the DLTs observed in each cohort. A DLT was defined as an adverse event (AE) (excluding anorexia and fatigue) or an abnormal laboratory value occurring within the first week (up to Week 2) following lanreotide PRF administration and during the entire study duration, assessed as unrelated to acromegaly, intercurrent illness or concomitant medications and which met any of the pre-established toxicity criteria. If no DLTs were reported then no MTD could be defined.
Time Frame: From Day 1 up to Week 25.
Population: The safety population was all subjects who received the single dose of lanreotide PRF and had at least one post baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
participants | 0 | 0 | 0

2. Primary Outcome: PK Analysis of Lanreotide: Maximum Observed Serum Concentration (Cmax).
Description: Blood samples for determination of lanreotide serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8,12 and 24 hours post-dose, on Days 3 and 5 and at Weeks 2, 3, 5, 9 and 13 after lanreotide PRF administration. Samples were also collected during follow-up at Weeks 17, 21 and 25 (or EW).
  Mean serum lanreotide Cmax values were determined using non-compartmental analysis.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: The PK valid population consisted of subjects who received at least 1 dose and had no major protocol deviations affecting the PK variables, and who had a sufficient number of serum lanreotide concentrations to estimate the main PK parameters. Only subjects with data available for analysis and who were not pre-treated with lanreotide are presented.
Measure: Mean (Standard Deviation); unit: nanograms/millilitre (ng/mL)
Groups:
- Lanreotide PK Set: 180 mg Lanreotide PRF: The lanreotide PK dataset included the 9 subjects from the PK valid population who were not pre-treated with lanreotide and who received 1 deep subcutaneous injection of 180 mg lanreotide PRF.
- Lanreotide PK Set: 270 mg Lanreotide PRF: The lanreotide PK dataset included the 7 subjects from the PK valid population who were not pre-treated with lanreotide and who received 1 deep subcutaneous injection of 270 mg lanreotide PRF. The 2 subjects previously treated with a stable dose of lanreotide Autogel were expected to have a detectable pre-dose concentration and it was considered relevant to exclude them.
- Lanreotide PK Set: 360 mg Lanreotide PRF: The lanreotide PK dataset included 6 subjects from the PK valid population who were not pre-treated with lanreotide and who received 1 deep subcutaneous injection of 360 mg lanreotide PRF. The 3 subjects previously treated with a stable dose of lanreotide Autogel were expected to have a detectable pre-dose concentration and it was considered relevant to exclude them.
Arm/Group | Lanreotide PK Set: 180 mg Lanreotide PRF | Lanreotide PK Set: 270 mg Lanreotide PRF | Lanreotide PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 7 | 6
nanograms/millilitre (ng/mL) | 19.0 (15.7) | 14.0 (10.3) | 20.5 (5.86)

3. Primary Outcome: PK Analysis of Lanreotide: Time to Reach Maximum Serum Concentration (Tmax).
Description: Blood samples for determination of lanreotide serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8,12 and 24 hours post-dose, on Days 3 and 5 and at Weeks 2, 3, 5, 9 and 13 after lanreotide PRF administration. Samples were also collected during follow-up at Weeks 17, 21 and 25 (or EW).
  Median serum lanreotide Tmax values were determined using non-compartmental analysis.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Groups:
- Lanreotide PK Set: 360 mg Lanreotide PRF: The lanreotide PK dataset included the 6 subjects from the PK valid population who were not pre-treated with lanreotide and who received 1 deep subcutaneous injection of 360 mg lanreotide PRF. The 3 subjects previously treated with a stable dose of lanreotide Autogel were expected to have a detectable pre-dose concentration and it was considered relevant to exclude them.
Arm/Group | Lanreotide PK Set: 180 mg Lanreotide PRF | Lanreotide PK Set: 270 mg Lanreotide PRF | Lanreotide PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 7 | 6
days | 0.250 [0.167 to 1.00] | 0.253 [0.167 to 1.00] | 0.250 [0.167 to 0.333]

4. Primary Outcome: PK Analysis of Lanreotide: Apparent Terminal Elimination Half-life (t1/2).
Description: Blood samples for determination of lanreotide serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8,12 and 24 hours post-dose, on Days 3 and 5 and at Weeks 2, 3, 5, 9 and 13 after lanreotide PRF administration. Samples were also collected during follow-up at Weeks 17, 21 and 25 (or EW).
  Mean serum lanreotide t1/2 values were determined using non-compartmental analysis. Only values fulfilling the determination rules for t1/2 were analysed.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lanreotide PK Set: 180 mg Lanreotide PRF | Lanreotide PK Set: 270 mg Lanreotide PRF | Lanreotide PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 7 | 5 | 4
days | 54.2 (17.0) | 61.7 (13.9) | 63.1 (13.3)

5. Primary Outcome: PK Analysis of Lanreotide: Area Under the Serum Concentration-time Curve From Time 0 to 85 Days (AUC0-85).
Description: Blood samples for determination of lanreotide serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8,12 and 24 hours post-dose, on Days 3 and 5 and at Weeks 2, 3, 5, 9 and 13 after lanreotide PRF administration. Sample were also collected during follow-up at Weeks 17, 21 and 25 (or EW).
  Mean serum lanreotide AUC0-85 values were determined using non-compartmental analysis.
Time Frame: From Baseline (pre-dose) up to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Lanreotide PK Set: 180 mg Lanreotide PRF | Lanreotide PK Set: 270 mg Lanreotide PRF | Lanreotide PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 7 | 6
ng*day/mL | 161 (97.6) | 179 (54.2) | 265 (87.1)

6. Primary Outcome: PK Analysis of Lanreotide: Area Under the Serum Concentration-time Curve Extrapolated to Infinity (AUC0-∞).
Description: Blood samples for determination of lanreotide serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8,12 and 24 hours post-dose, on Days 3 and 5 and at Weeks 2, 3, 5, 9 and 13 after lanreotide PRF administration. Samples were also collected during follow-up at Weeks 17, 21 and 25 (or EW).
  Mean serum lanreotide AUC0-∞ values were determined using non-compartmental analysis. Only values fulfilling the accuracy determination rules for AUC0-∞ were analysed.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Lanreotide PK Set: 180 mg Lanreotide PRF | Lanreotide PK Set: 270 mg Lanreotide PRF | Lanreotide PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 3 | 2 | 3
ng*day/mL | NA (NA) — When more than 1/3 of the values did not fulfil accuracy determination rules, the descriptive statistics were not calculated. | NA (NA) — When more than 1/3 of the values did not fulfil accuracy determination rules, the descriptive statistics were not calculated. | NA (NA) — When more than 1/3 of the values did not fulfil accuracy determination rules, the descriptive statistics were not calculated.

7. Secondary Outcome: Overall Summary of Number of Subjects With AEs.
Description: AEs reported by the investigators using the National Cancer Institute-Common Toxicity Criteria (NCI CTCAE) classification (Version 4.03) and incidence of all reported treatment emergent AEs (TEAEs) and serious AEs (SAEs) are presented by dose cohort. AEs were assigned to a NCI CTCAE Grade from 1 through 5 as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening or requiring hospitalisation; Grade 4: Life-threatening consequences; Grade 5: Death related to AE. TEAEs were defined as any AE that occurs during the active phase of the study (between the start of the 3 month treatment period and 3 months after the end of study treatment). The worst intensity of TEAES at each grade are reported for all and for related TEAES. In the event of multiple occurrences of the same AEs being reported by the same subject, the maximum intensity and the most serious causality were reported.
Time Frame: From Day -42 up to Week 25.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
participants
  TEAEs | 6 | 7 | 7
  Related TEAEs | 2 | 3 | 4
  TEAEs leading to study drug withdrawal | 0 | 0 | 0
  SAEs | 1 | 0 | 1
  Serious TEAEs | 1 | 0 | 1
  Serious related TEAEs | 0 | 0 | 0
  AEs leading to death | 0 | 0 | 0
  Worst TEAE: Grade 1 | 1 | 3 | 5
  Worst TEAE: Grade 2 | 3 | 4 | 1
  Worst TEAE: Grade 3 | 2 | 0 | 1
  Worst TEAE: Grade 4 | 0 | 0 | 0
  Worst TEAE: Grade 5 | 0 | 0 | 0
  Worst related TEAE: Grade 1 | 0 | 1 | 3
  Worst related TEAE: Grade 2 | 2 | 2 | 1
  Worst related TEAE: Grade 3 | 0 | 0 | 0
  Worst related TEAE: Grade 4 | 0 | 0 | 0
  Worst related TEAE: Grade 5 | 0 | 0 | 0

8. Secondary Outcome: PK Analysis of Glycofurol Excipients: Cmax.
Description: Blood samples for determination of the excipients (N1-glycofurol and N2-glycofurol) serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8, 12 and 24 hours post-dose and on Days 3 and 5. Mean serum N1-glycofurol and N2-glycofurol Cmax values were determined using non-compartmental analysis.
Time Frame: From Baseline (pre-dose) up to Day 5.
Population: The PK valid population consisted of subjects who received at least 1 dose and had no major protocol deviations affecting the PK variables, and who had a sufficient number of serum lanreotide concentrations to estimate the main PK parameters. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Glycofurol PK Set: 180 mg Lanreotide PRF: This glycofurol dataset included 9 subjects from the PK valid population who had a sufficient number of serum glycofurol concentrations to estimate the main glycofurol PK parameters (Cmax, Tmax, and AUC) and who received 1 deep subcutaneous injection of 180 mg lanreotide PRF.
- Glycofurol PK Set: 270 mg Lanreotide PRF: This glycofurol dataset included 9 subjects from the PK valid population who had a sufficient number of serum glycofurol concentrations to estimate the main glycofurol PK parameters (Cmax, Tmax, and AUC) and who received 1 deep subcutaneous injection of 270 mg lanreotide PRF.
- Glycofurol PK Set: 360 mg Lanreotide PRF: Due to bioanalytical issues, no results for the excipient N1-glycofurol and N2-glycofurol for this cohort were available at the time of the PK analysis.
Arm/Group | Glycofurol PK Set: 180 mg Lanreotide PRF | Glycofurol PK Set: 270 mg Lanreotide PRF | Glycofurol PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 0
ng/mL
  N1-glycofurol | 75.4 (65.6) | 61.7 (17.2) |
  N2-glycofurol | 79.7 (72.1) | 62.1 (18.4) |

9. Secondary Outcome: PK Analysis of Glycofurol Excipients: Tmax.
Description: Blood samples for determination of the excipients (N1-glycofurol and N2-glycofurol) serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8, 12 and 24 hours post-dose and on Days 3 and 5.
  Median serum N1-glycofurol and N2-glycofurol Tmax values were determined using non-compartmental analysis.
Time Frame: From Baseline (pre-dose) up to Day 5.
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Glycofurol PK Set: 180 mg Lanreotide PRF | Glycofurol PK Set: 270 mg Lanreotide PRF | Glycofurol PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 0
hours
  N1-glycofurol | 2.00 [1.00 to 3.92] | 2.00 [1.00 to 4.00] |
  N2-glycofurol | 2.00 [1.00 to 3.92] | 2.00 [1.00 to 4.00] |

10. Secondary Outcome: PK Analysis of Glycofurol Excipients: AUC0-∞ and Area Under the Serum Concentration Time Curve From Time 0 to Last Quantifiable Timepoint (AUC0-t).
Description: Blood samples for determination of the excipients (N1-glycofurol and N2-glycofurol) serum concentrations were collected at Baseline (pre-dose), at 1, 2, 4, 6, 8, 12 and 24 hours post-dose and on Days 3 and 5.
  Mean serum N1-glycofurol and N2-glycofurol AUC0-∞ and AUC0-t values were determined using non-compartmental analysis. Only AUC0-∞ values fulfilling the accuracy determination rules were analysed.
Time Frame: From Baseline (pre-dose) up to Day 5.
Population: The PK valid population consisted of subjects who received at least 1 dose and had no major protocol deviations affecting the PK variables, and who had a sufficient number of serum lanreotide concentrations to estimate the main PK parameters.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glycofurol PK Set: 180 mg Lanreotide PRF | Glycofurol PK Set: 270 mg Lanreotide PRF | Glycofurol PK Set: 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 0
ng*h/mL
  AUC0-∞: N1-glycofurol: number analyzed (Participants) | 8 | 8 | 0
  AUC0-∞: N1-glycofurol | 779 (205) | 1049 (195) |
  AUC0-∞: N2-glycofurol: number analyzed (Participants) | 8 | 8 | 0
  AUC0-∞: N2-glycofurol | 1008 (268) | 1359 (282) |
  AUC0-t: N1-glycofurol | 783 (193) | 1082 (238) |
  AUC0-t: N2-glycofurol | 1007 (257) | 1360 (285) |

11. Secondary Outcome: PD Analysis: Mean Change From Baseline in Insulin-like Growth Factor 1 (IGF-1).
Description: Blood samples were collected for the determination of IGF-1 in serum at Baseline (pre-dose), 6 hours post-dose and at Weeks 5, 9 and 13. Samples were also collected during follow-up at Weeks 17, 21 and 25 (or EW). Serum concentrations of IGF-1 were calculated using the Immulite 2000 Platform for all subjects in the safety population. The production of the reagent kits was stopped by the vendor during the study. The old reagent kits were used for Cohorts 1 and 2 until their expiry date and then the kits were switched to a new reagent and used for remaining subjects in Cohorts 2 and 3. Summary data for serum concentrations of IGF-1 were obtained using both methods (old and new reagent) and the mean change from Baseline at each time point is presented.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: The safety population was all subjects who received the single dose of lanreotide PRF and had at least one post baseline safety assessment. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
ng/mL
  Old Reagent: 6 hours post-dose: number analyzed (Participants) | 9 | 8 | 4
  Old Reagent: 6 hours post-dose | -1.8 (18.9) | -7.1 (17.2) | -46.5 (46.7)
  Old Reagent: Week 5: number analyzed (Participants) | 9 | 9 | 2
  Old Reagent: Week 5 | 2.4 (41.3) | 27.9 (32.8) | -32.0 (49.5)
  Old Reagent: Week 9: number analyzed (Participants) | 9 | 9 | 0
  Old Reagent: Week 9 | 72.3 (61.3) | 71.4 (72.7) |
  Old Reagent: Week 13: number analyzed (Participants) | 7 | 9 | 0
  Old Reagent: Week 13 | 53.4 (67.9) | 111.1 (129.3) |
  Old Reagent: Week 17: number analyzed (Participants) | 7 | 6 | 0
  Old Reagent: Week 17 | 48.3 (62.7) | 96.2 (43.8) |
  Old Reagent: Week 21: number analyzed (Participants) | 5 | 4 | 0
  Old Reagent: Week 21 | 72.4 (84.4) | 135.5 (80.5) |
  Old Reagent: Week 25 (EOS/EW): number analyzed (Participants) | 9 | 9 | 0
  Old Reagent: Week 25 (EOS/EW) | 86.3 (81.4) | 136.4 (83.5) |
  New Reagent: 6 hours post-dose: number analyzed (Participants) | 0 | 2 | 9
  New Reagent: 6 hours post-dose |  | 6.0 (5.7) | -11.6 (15.9)
  New Reagent: Week 5: number analyzed (Participants) | 0 | 2 | 10
  New Reagent: Week 5 |  | 3.0 (8.5) | 1.3 (38.4)
  New Reagent: Week 9: number analyzed (Participants) | 0 | 2 | 9
  New Reagent: Week 9 |  | 13.0 (9.9) | 25.2 (33.6)
  New Reagent: Week 13: number analyzed (Participants) | 0 | 2 | 10
  New Reagent: Week 13 |  | 30.0 (43.8) | 47.1 (43.9)
  New Reagent: Week 17: number analyzed (Participants) | 0 | 2 | 8
  New Reagent: Week 17 |  | 20.5 (17.7) | 40.9 (46.8)
  New Reagent: Week 21: number analyzed (Participants) | 0 | 2 | 7
  New Reagent: Week 21 |  | 65.0 (58.0) | 56.9 (35.6)
  New Reagent: Week 25 (EOS/EW): number analyzed (Participants) | 0 | 2 | 10
  New Reagent: Week 25 (EOS/EW) |  | 45.5 (17.7) | 64.1 (68.0)

12. Secondary Outcome: PD Analysis: Mean Change From Baseline in Growth Hormone (GH).
Description: GH cycle assessments were performed by taking 5 samples in the morning (with a sample taken every 30 minutes for 2 hours) at Baseline (pre-dose), Week 5 and Week 13. Summary data for the mean of the 5 samplings of the GH cycle were generated and the mean change from Baseline at each time point is presented.
Time Frame: From Baseline (pre-dose) up to Week 13.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
ng/mL
  Week 5 | 0.268 (0.344) | 0.367 (0.926) | -0.228 (0.777)
  Week 13: number analyzed (Participants) | 7 | 9 | 10
  Week 13 | 0.667 (0.473) | 0.684 (0.863) | 0.003 (1.761)

13. Secondary Outcome: PD Analysis: Mean Change From Baseline in Free Triiodothyroxine (FT3) and Free Thyroxine (FT4).
Description: Blood samples were collected for the determination of FT3 and FT4 in serum at Baseline (pre-dose) and at Weeks 2, 5, 13 and 25 (or EW). Summary data for serum concentrations of FT3 and FT4 were calculated and the mean change from Baseline at each time point is presented.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: picomole/litre (L)
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
picomole/litre (L)
  FT3: Week 2: number analyzed (Participants) | 9 | 9 | 9
  FT3: Week 2 | -0.278 (0.518) | -0.164 (0.517) | -0.374 (0.479)
  FT3: Week 5: number analyzed (Participants) | 9 | 9 | 9
  FT3: Week 5 | -0.132 (0.429) | -0.170 (0.705) | 0.170 (0.452)
  FT3: Week 13: number analyzed (Participants) | 7 | 9 | 10
  FT3: Week 13 | 0.100 (0.590) | 0.191 (0.912) | 0.438 (0.481)
  FT3: Week 25 (EOS/EW) | 0.268 (0.388) | 0.295 (0.626) | 0.396 (0.684)
  FT4: Week 2: number analyzed (Participants) | 9 | 9 | 9
  FT4: Week 2 | 0.50 (1.58) | -0.02 (1.43) | -0.68 (1.07)
  FT4: Week 5: number analyzed (Participants) | 9 | 9 | 9
  FT4: Week 5 | 1.18 (2.31) | 0.33 (2.52) | -0.67 (2.19)
  FT4: Week 13: number analyzed (Participants) | 7 | 9 | 10
  FT4: Week 13 | 1.69 (2.16) | 1.80 (3.59) | -0.46 (1.39)
  FT4: Week 25 (EOS/EW): number analyzed (Participants) | 9 | 8 | 10
  FT4: Week 25 (EOS/EW) | 0.81 (2.55) | 1.06 (2.39) | 0.38 (2.03)

14. Secondary Outcome: PD Analysis: Mean Change From Baseline in Thyroid Stimulating Hormone (TSH).
Description: Blood samples were collected for the determination of TSH in serum at Baseline (pre-dose) and at Weeks 2, 5, 13 and 25 (or EW). Summary data for serum concentrations of TSH were calculated and the mean change from Baseline at each time point is presented.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
mIU/L
  Week 2: number analyzed (Participants) | 9 | 9 | 9
  Week 2 | -0.222 (0.562) | 0.119 (0.315) | 0.047 (0.844)
  Week 5: number analyzed (Participants) | 9 | 9 | 9
  Week 5 | -0.156 (0.577) | 0.062 (0.670) | 0.051 (0.534)
  Week 13: number analyzed (Participants) | 7 | 9 | 10
  Week 13 | -0.404 (0.710) | -0.060 (0.897) | 0.601 (1.080)
  Week 25 (EOS/EW): number analyzed (Participants) | 9 | 8 | 10
  Week 25 (EOS/EW) | -0.480 (0.593) | 0.073 (0.450) | 0.235 (0.671)

15. Secondary Outcome: PD Analysis: Mean Change From Baseline in Prolactin.
Description: Blood samples were collected for the determination of prolactin in serum at Baseline (pre-dose) and at Weeks 2, 5, 13 and 25 (or EW). Summary data for serum concentration of prolactin were calculated and the mean change from Baseline at each time point is presented.
Time Frame: From Baseline (pre-dose) up to Week 25.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
Number analyzed (Participants) | 9 | 9 | 10
mU/L
  Week 2: number analyzed (Participants) | 9 | 9 | 9
  Week 2 | -33.2 (54.9) | 37.6 (36.1) | 1.0 (49.3)
  Week 5: number analyzed (Participants) | 9 | 9 | 9
  Week 5 | -10.4 (53.2) | 16.3 (81.2) | 0.3 (50.7)
  Week 13: number analyzed (Participants) | 7 | 9 | 10
  Week 13 | -1.9 (66.5) | 33.9 (78.5) | -6.4 (47.1)
  Week 25 (EOS/EW): number analyzed (Participants) | 9 | 8 | 10
  Week 25 (EOS/EW) | 19.3 (53.5) | 58.3 (86.6) | -3.1 (55.9)

ADVERSE EVENTS:
Time Frame: Each subject was assessed for TEAEs over an approximate 6 month period. TEAEs were collected over the 32 month study duration.
Description: TEAES were monitored for the safety population which was defined as all subjects who received the single dose of lanreotide PRF and had at least one post baseline safety assessment.
Arm/Group | 180 mg Lanreotide PRF | 270 mg Lanreotide PRF | 360 mg Lanreotide PRF
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 6/9 | 7/9 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg Lanreotide PRF (N=9) | 270 mg Lanreotide PRF (N=9) | 360 mg Lanreotide PRF (N=10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg Lanreotide PRF (N=9) | 270 mg Lanreotide PRF (N=9) | 360 mg Lanreotide PRF (N=10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (2)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection Site Haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection Site Induration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection Site Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Conjunctival Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
No glycofurol excipient PK results are available for 360mg Lanreotide PRF at this time. A total of 28 subjects were allowed to enrol rather than the 27 subjects planned as it was considered unethical not to enrol a consented eligible subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT02396953/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02396953/SAP_001.pdf